CLINICAL TRIAL: NCT00555061
Title: An Open-Label, Non-Comparative Study to Assess the Pharmacokinetics, Safety and Efficacy of Topical Retapamulin (SB-275833) Ointment, 1%, Twice Daily for Five Days in the Treatment of Uncomplicated Skin and Skin Structure Infections in Pediatric Subjects Aged 2 to 24 Months
Brief Title: Pharmacokinetics of Retapamulin in Pediatric Subjects With Uncomplicated Skin Infections.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOC106489
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Results first posted 2010-04-30 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Skin Infections, Bacterial
Keywords: SID; impetigo; pharmacokinetics; Retapamulin ointment, 1%; Skin abnormalities; Dermatoses; pediatric; infection; SITL
MeSH Terms: conditions — Cellulitis; Sudden Infant Death; Impetigo; Skin Abnormalities; Skin Diseases; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Single Arm Retapamulin 1% Ointment
  Interventions: Drug: Retapamulin Ointment, 1%

INTERVENTIONS:
Drug: Retapamulin Ointment, 1% — 1% Ointment
  Other Names: Retapamulin Ointment; 1%

SUMMARY:
A study to evaluate the pharmacokinetics of Retapamulin Ointment, 1%, in pediatric subjects (2-24 months) with secondarily-infected traumatic lesions, secondarily-infected dermatoses, or impetigo (bullous and non-bullous).

ELIGIBILITY:
Inclusion criteria:

* Subject Age: The subject is ≥2 months to ≤24 months of age at study entry
* Subject Diagnosis: The subject has a diagnosis of secondarily-infected traumatic lesion (SITL), secondarily-infected dermatoses (SID), or primary impetigo (bullous or non-bullous) that is suitable for treatment with topical antibacterial therapy:

The subject has a small laceration, sutured wound or abrasion, which has a secondary bacterial infection. The infected portion of the laceration or sutured wound should not exceed 10cm in length with surrounding erythema not extending more than 2cm from the edge of the wound. Abrasions should not exceed 2% of the total body surface area with surrounding erythema not extending more than 2cm from the edge of the abrasion.

The subject has a diagnosis of inflammatory skin disease (i.e., dermatosis), such as atopic dermatitis or contact dermatitis, which has a secondary bacterial infection. The infected portion of the lesion(s) should not exceed 2% of the total body surface area.

Impetigo: The subject has a lesion or group of £10 discrete localized lesions on otherwise healthy skin, characterized by red spots or blisters without crusts which later progress to lesions which ooze and form yellow or honey-colored crusts surrounded by an erythematous margin.

* Subject SIRS Score: The subject has a total SIRS score of at least 8 (Appendix 1 Skin Infection Rating Scale)
* Protocol Compliance: The parent/legal guardian is willing to comply with the protocol
* Informed Consent: The parent/legal guardian has given written informed, dated consent for the subject to participate in the study
* French Subjects: In France, a subject will be eligible for inclusion in this study if either affiliated to or a beneficiary of a social security category

Exclusion criteria:

* The subject has demonstrated a previous hypersensitivity reaction to pleuromutilin or any component of the ointment (refer to the Investigator Brochure for composition of Retapamulin ointment, 1%)
* The subject was considered to be premature at birth (<37 weeks gestation)
* The subject has a secondarily-infected animal/human bite, or a puncture wound
* The subject has an abscess
* The subject has a chronic ulcerative lesion that is unlikely to have Staphylococcus aureus or Streptococcus pyogenes as the causative agent
* The subject has systemic signs and symptoms of infection (such as fever; defined as a temperature equivalent to a rectal temperature greater than 101°F or 38.3°C)
* The subject has a bacterial skin infection which, due to area, depth or severity, in the opinion of the investigator, cannot be appropriately treated by a topical antibiotic
* The subject has more than one type of infected lesion as defined in the protocol
* The subject requires surgical intervention for treatment of the infection prior to enrollment in the study, or is likely to require such intervention during the course of the study
* The subject has applied any topical therapeutic agent (including glucocorticoid steroids, antibacterials or antifungals) directly to the infected wound/lesion, within 24 hours prior to study entry
* The subject has received one or more days of treatment with a systemic antibacterial within 72 hours of study entry
* The subject is receiving systemic corticosteroids at a dose of >0.125mg/kg per day of prednisone (or the equivalent)
* The subject has a known, pre-existing, serious underlying disease that could be imminently life-threatening
* The subject has participated in any study using an investigational drug during the previous 30 days prior to entering the study
* The subject has been previously enrolled in this study or in any other study involving Retapamulin

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (6):
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Bentonville, Arkansas
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Woburn, Massachusetts
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- GSK Investigational Site, San José, Costa Rica
- Germany (5):
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
- GSK Investigational Site, México, Mexico
- Netherlands (6):
  - GSK Investigational Site, Alphen aan den Rijn
  - GSK Investigational Site, Losser
  - GSK Investigational Site, Roelofarendsveen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Soerendonk
  - GSK Investigational Site, Woerden
- South Africa (2):
  - GSK Investigational Site, Benoni
  - GSK Investigational Site, Newtown
- GSK Investigational Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: TOC106489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: TOC106489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TOC106489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: TOC106489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: TOC106489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: TOC106489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TOC106489 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Retapamulin Ointment, 1%: Retapamulin ointment, 1%, administered twice daily for 5 consecutive days
Period: Overall Study
Arm/Group | Retapamulin Ointment, 1%
Started | 87 (One participant did not receive study medication and was not included in the analysis population.)
Completed | 78
Not Completed | 9
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — Participant enrolled, but never treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Retapamulin Ointment, 1%
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: months] — One participant was enrolled, but was withdrawn prior to assessments and did not receive study medication; therefore, this participant was not included in the study population.
  months | 10.6 (6.89)
Gender [Count of Participants; unit: Participants] — One participant was enrolled, but was withdrawn prior to assessments and did not receive study medication; therefore, this participant was not included in the study population.
  Participants
    Female | 32
    Male | 54
Race/Ethnicity, Customized [Number; unit: participants] — One participant was enrolled, but was withdrawn prior to assessments and did not receive study medication; therefore, this participant was not included in the study population.
  participants
    African American/African Heritage | 46
    White/Caucasian | 36
    American Indian or Alaska Native | 1
    Central/South Asian | 1
    East Asian | 1
    Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Measurable Plasma Concentrations, by Age Group
Description: Pharmacokinetic (PK) samples were collected randomly in the window of 4 to 8 hours post-dose (except one at 3 hours and one at 11 hours post-dose) after the first daily dose of treatment on Day 3 or Day 4. The lower limit of quantification (LLQ) for retapamulin was 0.5 ng/mL.
Time Frame: Days 3 to 4; 4 to 8 hours post-dose of the first dose of the day
Population: Pharmacokinetic (PK) Population: all participants who received at least one dose of study medication and who had PK samples taken. Seven participants did not have PK samples collected.
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment, 1%
Number analyzed (Participants) | 79
participants
  All ages | 36
  ≥2 months to ≤6 months | 17
  >6 months to ≤12 months | 10
  >12 months to ≤24 months | 9

2. Secondary Outcome: Number of Participants With Clinical Success at Follow-up, by Type of Skin Infection and by Age
Description: SID = Secondarily Infected Dermatoses; SITL = Secondarily Infected Traumatic Lesions. Clinical Success is the number of participants with resolution of signs/symptoms of infection or improvement such that no additional antibiotic therapy was needed.
Time Frame: Follow-up, Days 12 to 16
Population: Intent-to-Treat Clinical (ITTC) Population: all participants who received at least one dose of study medication; the number of participants who were clinical successes out of the total number in each respective category is shown
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment, 1%
Number analyzed (Participants) | 86
participants
  Impetigo, ≥2 months to ≤6 months, n=11 | 10
  Impetigo, >6 months to ≤12 months, n=18 | 17
  Impetigo, >12 months to ≤24 months, n=18 | 17
  SID, ≥2 months to ≤6 months, n=17 | 11
  SID, >6 months to ≤12 months, n=9 | 7
  SID, >12 months to ≤24 months, n=4 | 4
  SITL, ≥2 months to ≤6 months, n=1 | 1
  SITL, >6 months to ≤12 months, n=2 | 2
  SITL, >12 months to ≤24 months, n=6 | 6

3. Secondary Outcome: Bacteriological Success Rate at Follow-up, by Baseline Pathogen
Description: Bacteriological success is defined as: (1) Bacteriological Eradication, elimination of the baseline pathogen via culture results; (2) Presumed Bacteriological Eradication, clinical success plus no culturable material from the wound; or (3) Colonization, new pathogen identified at Follow-up in a non-symptomatic participant who does not require additional antibiotic therapy. The number of pathogens eradicated out of the number isolated (shown as "n" in the category title) for each respective category is shown.
Time Frame: Follow-up, Days 12 to 16
Population: ITTB (Intent-to-Treat Bacteriological) Population: participants who had at least one dose of study medication and a clinical diagnosis of infection plus a pathogen isolated at Baseline. Participants with more than one pathogen may be represented in the table more than once.
Measure: Number; unit: number of pathogens eradicated
Arm/Group | Retapamulin Ointment, 1%
Number analyzed (Participants) | 61
number of pathogens eradicated
  All pathogens, n=93 | 79
  Staphylococcus aureus (SA), n=44 | 40
  Methicillin-resistant SA, n=3 | 3
  Methicillin-susceptible SA, n=41 | 37
  Mupirocin-susceptible SA, n=44 | 40
  Fuscidic acid-resistant SA, n=2 | 2
  Fuscidic acid-susceptible SA, n=42 | 38
  Streptococcus pyogenes, n=9 | 9
  Other Gram (+) pathogens, n=11 | 9
  Gram (-) pathogens, n=29 | 21

4. Secondary Outcome: Number of Participants by Age With Therapeutic Response of Success
Description: Therapeutic response is a measure of the overall efficacy response; a response of "therapeutic success" was based on both clinical success and bacteriological success in a given participant.
Time Frame: Follow-up, Days 12 to 16
Population: ITTB and ITTC Populations. The number analyzed is the number of participants who were clinical successes both in the ITTC Population and the ITTB Population; the number of participants who were therapeutic successes out of the total number in each respective category is shown.
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment, 1%
Number analyzed (Participants) | 61
participants
  All ages | 51
  >2 months to <=6 months, n=21 | 15
  >6 months to <=12 months, n=20 | 17
  >12 months to <=24 months, n=20 | 19

ADVERSE EVENTS:
Arm/Group | Retapamulin Ointment, 1%
Serious Adverse Events (participants affected / at risk) | 1
Other Adverse Events (participants affected / at risk) | 11
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Retapamulin Ointment, 1%
Cough (Respiratory, thoracic and mediastinal disorders) | 1/86
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Retapamulin Ointment, 1%
Diarrhea (Gastrointestinal disorders) | 2/86
Atopic dermatitis (Skin and subcutaneous tissue disorders) | 2/86
Influenza (Infections and infestations) | 2/86
Abdominal pain (Gastrointestinal disorders) | 1/86
Vomiting (Gastrointestinal disorders) | 1/86
Dermatitis (Skin and subcutaneous tissue disorders) | 1/86
Impetigo (Infections and infestations) | 1/86
Skin fissure (Skin and subcutaneous tissue disorders) | 1/86
Hypersensitivity (Immune system disorders) | 1/86
Pharyngitis (Infections and infestations) | 1/86
Hypochromic anemia (Blood and lymphatic system disorders) | 1/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.